CLINICAL TRIAL: NCT02445495
Title: A Single Centre Retrospective Chart Review Study to Assess the Efficacy of the GenesisPlus 1064 nm Nd:YAG Laser in the Treatment of Onychomycosis
Brief Title: Chart Review of the Efficacy of the GenesisPlus 1064 nm Nd:YAG Laser in the Treatment of Onychomycosis
Status: Completed | Type: Observational
Sponsor: Jason K Rivers, MD, FRCPC, FAAD (Other)
Collaborators: Cutera Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jason K Rivers, MD, FRCPC, FAAD, Principal Investigator, Pacific Dermaesthetics
Organization: Pacific Dermaesthetics (Other)
Other Study IDs: PDA288
Record Dates: First submitted 2015-04-30; First posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: GenesisPlus 1064 nm Nd:YAG laser — Genesis Plus 1064 nm Nd: YAG laser to treat onychomycosis
  Other Names: Cutera®

SUMMARY:
The purpose of this study is to determine if toenail onychomycosis can be reduced by means of exposure to laser energy from the Cutera® GenesisPlus 1064 Nd:YAG laser system.

DETAILED DESCRIPTION:
This is a retrospective, open-label, single-centre study for the collection of clinical data on the efficacy and safety of the Cutera® GenesisPlus 1064 nm Nd:YAG laser for the treatment of nail fungus (onychomycosis). Safety and efficacy of treatment with the GenesisPlus laser will be evaluated by (1) assessment of subject's great toenail photographs at baseline and after two treatments with GenesisPlus Laser utilizing planimetry measurement of infected vs. clear nail area in target toenail photographs, (2) by clinical and subjective review of acute and follow up adverse events that may have resulted from laser treatment of the target toenails.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects, age 18 to 80 years (inclusive).
2. Subject with a clinical diagnosis of onychomycosis of one or both great toenails at baseline.
3. Subject with a positive potassium hydroxide (KOH) stain and/or fungal culture.
4. Subject has baseline and post treatment digital photographs of target great toenails.
5. Subjects provided informed consent for treatment of nails with the Cutera GenesisPlus laser system.

Exclusion Criteria:

1. Subjects have received laser treatment of the infected great toenail(s) with a non-Cutera® laser system within twelve (12) months prior to Cutera® GenesisPlus laser treatment.
2. Subjects have had a history or clinical diagnosis of moccasin type tinea pedis, lichen planus, psoriasis or bacterial nail infection.
3. Subjects had a history or clinical diagnosis of coexisting disorders that may potentially demonstrate nail manifestations.
4. Systemic antifungal medication within six (6) months prior to or following Cutera® GenesisPlus laser treatment.
5. Subjects who have had a history or clinical diagnosis of repetitive nail trauma prior to treatment.
6. Subjects who have participated in any clinical research study within thirty (30) days prior to or within 210 days following final Cutera® GenesisPlus laser treatment.
7. Subjects who were pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 participants at primary clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
change in % of infected toenail involvement | change from baseline up to 6 months
  onychomycosis involvement